CLINICAL TRIAL: NCT02197130
Title: A Phase 2, Randomized, Placebo Controlled, Double Blind Proof-of-concept Study Of The Efficacy And Safety Of Pf-02545920 In Subjects With Huntington's Disease
Brief Title: Randomized, Placebo Controlled Study Of The Efficacy And Safety Of PF-02545920 In Subjects With Huntington's Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: A8241021; 2014-001291-56 (EudraCT Number)
Record Dates: First submitted 2014-07-16; First posted 2014-07-22 (Estimated); Results first posted 2017-11-17 (Actual); Last update posted 2017-11-17 (Actual); Status verified 2017-10

CONDITIONS: Huntington's Disease
Keywords: Huntington; chorea; total motor score; CAG repeat: total functional capacity; motor cognitive and behavioral symptoms
MeSH Terms: conditions — Huntington Disease; Chorea; Behavioral Symptoms | interventions — 2-((4-(1-methyl-4-pyridin-4-yl-1H-pyrazol-3-yl)phenoxy)methyl)quinoline

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 20 mg PF-02545920 BID (Experimental): 20 mg PF-02545920 BID
  Interventions: Drug: PF-02545920
- 5 mg PF-02545920 BID (Experimental): 5 mg PF-02545920 BID
  Interventions: Drug: PF-02545920
- Placebo BID (Placebo Comparator): Matching placebo
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: PF-02545920 — 20 mg twice a day (BID) for 26 weeks. Each 20 mg dose will be taken as 4 tablets of 5 mg. The 20mg dose will be titrated as follow: 5mg BID for 7 days, 10mg BID for 7 days, 15 mg BID for 7 days and 20 mg BID to week 26. Study drug will be provided in weekly blister cards.
  Arms: 20 mg PF-02545920 BID
Drug: PF-02545920 — 5 mg twice a day (BID) for 26 weeks. Each 5 mg dose will be taken as 4 tablets: one tablet of 5 mg and 3 tablets of matching placebo. The 5mg dose will not be titrated. Study drug will be provided in weekly blister cards.
  Arms: 5 mg PF-02545920 BID
Other: Placebo — Matching Placebo twice a day (BID) for 26 weeks. Each placebo dose will be taken as 4 tablets of matching Placebo. The placebo dose will not be titrated. Matching placebo will be provided in weekly blister cards.
  Arms: Placebo BID

SUMMARY:
This study is a 26 week, randomized, parallel group, double blind comparison of PF-02545920 5 mg, PF-02545920 20 mg, and placebo dosed BID in the treatment of motor impairment of subjects with Huntington's Disease. A total of approximately 260 subjects are planned to be randomized in the study. Primary endpoint is the change from baseline in the Total Motor Score (TMS) assessment of the Unified Huntington Disease Rating Scale (UHDRS) after 26 weeks of treatment. secondary endpoints will include change from baseline in the Total Maximum Chorea (TMC) score of the UHDRS after 13 and 26 weeks of treatment and Clinical Global Impression-Improvement score after 13 and 26 weeks of treatment.

ELIGIBILITY:
Inclusion Criteria:

* CAG repeat equal or greater than 36;
* Total motor score equal or greater than 10;
* Total functional capacity equal or greater than 7.

Exclusion Criteria:

* Clinically significant neurologic disorder other than Huntington's disease;
* Other severe acute psychiatric conditions, mania and/or psychosis;
* History of neutropenia, and myeloproliferative disorders;

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 272 (Actual)
Dates: Start 2014-09 (Actual); Primary Completion 2016-09 (Actual); Study Completion 2016-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (57):
- United States (22):
  - The Kirklin Clinic of UAB Hospital, Birmingham, Alabama
  - The University of Alabama at Birmingham, Birmingham, Alabama
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Mayo Clinic Arizona, Phoenix, Arizona
  - Mayo Clinic Arizona, Scottsdale, Arizona
  - University of California, Irvine, Irvine, California
  - Ronald Regan UCLA Medical Center Drug Information Center, Los Angeles, California
  - UCLA Neurology Clinic, Los Angeles, California
  - UCLA Radiology, Los Angeles, California
  - Rocky Mountain Movement Disorders Center, Englewood, Colorado
  - University of Florida Center for Movement Disorders and Neurorestoration, Gainesville, Florida
  - Indiana University Health Neuroscience Center, Indianapolis, Indiana
  - Massachusetts General Hospital, Charlestown, Massachusetts
  - Washington University School of Medicine, St Louis, Missouri
  - Albany Medical College, Albany, New York
  - Wake Forest Baptist Medical Center - Dept. of Neurology, Winston-Salem, North Carolina
  - Cleveland Clinic Foundation Hospital Pharmacy, Cleveland, Ohio
  - The Cleveland Clinic Foundation, Cleveland, Ohio
  - Davis Medical Center, Columbus, Ohio
  - The Wexner Medical Center at the Ohio State University, Columbus, Ohio
  - Wexner Medical Center at the Ohio State University, Columbus, Ohio
  - Baylor College of Medicine, Houston, Texas
- Canada (4):
  - The Centre for Huntington Disease, Vancouver, British Columbia
  - Centre for Movement Disorders, Toronto, Ontario
  - CHUM-Notre-Dame Hospital, Montreal, Quebec
  - CHUM Notre Dame, Pharmacie, Montreal, Quebec
- Germany (12):
  - Technische Universität München, München, Bavaria
  - Uniklinik RWTH Aachen, Aachen
  - Charite - Universitatsmedizin Berlin, Berlin
  - Prof. Dr. Carsten Saft, Bochum
  - Friedrich-Alexander-Universität, Erlangen
  - Prof. Dr. med. Stephan Klebe, Freiburg im Breisgau
  - Universitat zu Lubeck, Lübeck
  - Philipps Universitat Marburg, Marburg
  - George Huntington Institut, Münster
  - Kbo-Isar-Amper-Klinikum gGmbH, Taufkirchen
  - Universitätsklinikum Ulm, Ulm
  - Universitatsklinikum Wuerzburg, Würzburg
- Poland (4):
  - Copernicus Podmiot Leczniczy sp. z o.o., Gdansk
  - Krakowska Akademia Neurologii Sp. z o.o., Krakow
  - Solumed Centrum Medyczne, Poznan
  - Instytut Psychiatrii i Neurologii, Warsaw
- United Kingdom (15):
  - NHS Grampian, Clinical Genetics Centre, Aberdeen, Aberdeenshire
  - University Hospital Southampton NHS Foundation Trust, Southampton, Hampshire
  - Oxford University Hospitals NHS Trust, Oxford, Oxfordshire
  - Sheffield Teaching Hospitals NHS Foundation Trust, Sheffield, South Yorkshire
  - Birmingham & Solihull Mental Health NHS Foundation Trust, Birmingham, West Midlands
  - John Van Geest Centre for Brain Repair, Cambridge
  - University of Wales Hospital, Cardiff
  - NHS Greater Glasgow and Clyde, Glasgow
  - Clinical Research Facility, London
  - University College London Hospitals Huntington's Disease Research Centre, London
  - University College London Hospitals NHS Foundation Trust, London
  - Central Manchester University Hospitals NHS Foundation Trust, Manchester
  - The National Institute for Health Research/Wellcome Trust Clinical Research Facility, Manchester
  - St Nicholas Hospital, Newcastle upon Tyne
  - Newcastle Magnetic Resonance Centre, Newcastle upon Tyne

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A8241021

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 272 subjects (133 males and 139 females) were randomized and assigned study treatment.
Groups:
- PF-02545920 5 mg BID: Participants took 4 tablets packaged in blister packs (3 placebo tablets and one 5 mg PF-02545920) twice a day approximately every 12 hours from Baseline Day 1 (V2) to Week 26 (V9), at approximately the same time of day throughout the study. Study medication was swallowed whole, and was not manipulated or chewed prior to swallowing.
- Placebo: Participants took 4 tablets of placebo packaged in blister packs twice a day approximately every 12 hours, at approximately the same time of day throughout the study. Study medication was swallowed whole, and was not manipulated or chewed prior to swallowing.
- PF-02545920 20 mg BID: The 20 mg BID dose of PF-02545920 was titrated as follows: 5 mg BID for 7 days, 10 mg BID for 7 days, 15 mg BID for 7 days, then 20 mg BID for the remainder of the treatment phase. Participants took 4 tablets packaged in blister packs twice a day approximately every 12 hours, at approximately the same time of day throughout the study. The blister packs contained 3 placebo tablets and one 5 mg PF-02545920 tablet for Days 1-7, 2 placebo tablets and two 5 mg PF-02545920 tablets for Days 8-14, 1 placebo tablet and three 5 mg PF-02545920 tablets for Days 15-21, and four 5 mg PF-02545920 tablets from Day 22 through Day 182. Study medication was swallowed whole, and was not manipulated or chewed prior to swallowing.
Period: Overall Study
Arm/Group | PF-02545920 5 mg BID | Placebo | PF-02545920 20 mg BID
Started | 95 | 89 | 88
Received Treatment | 95 | 88 | 87
Completed | 79 | 81 | 56
Not Completed | 16 | 8 | 32
Not completed — Adverse Event | 13 | 4 | 23
Not completed — Death | 0 | 1 | 0
Not completed — Lost to Follow-up | 2 | 0 | 1
Not completed — Does not meet entrance criteria | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 3 | 4
Not completed — Other | 1 | 0 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | PF-02545920 5 mg BID | Placebo | PF-02545920 20 mg BID | Total
Number analyzed (Participants) | 95 | 88 | 87 | 270
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.3 (8.6) | 50.2 (9.4) | 48.4 (9.2) | 48.9 (9.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 42 | 54 | 43 | 139
  Male | 53 | 34 | 44 | 131

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in the Total Motor Score (TMS) Assessment of the Unified Huntington Disease Rating Scale (UHDRS) After 26 Weeks of Treatment.
Description: The UHDRS was a clinical rating scale which has been developed by the Huntington Disease Study Group (HSG) to provide a uniform assessment of the clinical features and course of Huntington's Disease (HD). The components of the full UHDRS assess motor function, cognition, behavior and functional abilities. The total motor score (TMS) assessed motor features of HD with standardized ratings of oculomotor function, dysarthria, chorea, dystonia, gait, and postural stability. Some items (such as chorea and dystonia) required grading each extremity (face, bucco-oral-lingual, and trunk) separately. Eye movements require both horizontal and vertical grades. The total motor impairment scores was the sum of all the individual 31 motor sub-items (each rated from 0 to 4), with higher scores indicating more severe motor impairment than lower scores. The range of TMS is 0-124.
Time Frame: Baseline, Week 26
Population: All participants who have been randomized and have taken at least one dose of PF-02545920 or placebo. Participants without post-dose measurements did not contribute to the analysis, except in the description of the baseline values.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | PF-02545920 20 mg BID | PF-02545920 5 mg BID | Placebo
Number analyzed (Participants) | 59 | 83 | 80
units on a scale | 0.4 (8.63) | -0.8 (7.30) | -1.4 (6.67)
Statistical Analysis 1: Comparison: PF-02545920 20 mg BID vs Placebo; Test type: Superiority or Other; p = 0.2033, MMRM; MMRM: A linear mixed-effect repeated measures model; Mean Difference (Net) = 1.52, 90% CI 2-sided [-0.45 to 3.49], Standard Error of Mean 1.192
Statistical Analysis 2: Comparison: PF-02545920 5 mg BID vs Placebo; Test type: Superiority or Other; p = 0.7549, MMRM; Mean Difference (Net) = -0.35, 90% CI 2-sided [-2.20 to 1.50], Standard Error of Mean 1.118

2. Secondary Outcome: Number of Participants That Met White Blood Count (WBC) and Absolute Neutrophil Count (ANC) Stopping Criteria
Description: The criteria for temporary study suspension was as follow: Criterion A: WBC count <=3000 cells/mm3 but >= 2000 cells/mm3 or ANC <= 1500 cells/mm3 but >= 1000 cells/mm3; Criterion B: WBC <= 2000 cells/mm3 or ANC <= 1000 cells/mm3; Criterion C: participants who are discontinued or permanently suspended due to WBC or ANC findings; Criterion D: ANC <= 500 cells/mm3
Time Frame: Screening, Day 1, 7, 14, 28, 56, 91, 133, 182 and follow-up visits (from Day 189 to 192)
Population: All participants with at least one dose of study medication.
Measure: Number; unit: participants
Arm/Group | PF-02545920 20 mg BID | PF-02545920 5 mg BID | Placebo
Number analyzed (Participants) | 87 | 95 | 88
participants
  Criterion A | 0 (8.63) | 1 (7.30) | 0 (6.67)
  Criterion B | 0 | 0 | 0
  Criterion C | 0 | 0 | 0
  Criterion D | 0 | 0 | 0

3. Secondary Outcome: Number of Participants With Adverse Events
Description: Adverse event (AE) was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship.
Time Frame: Day 1, 7, 14, 28, 56, 91, 133, 182 and follow-up visits (from Day 189 to 192)
Population: All participants with at least one dose of study medication.
Measure: Number; unit: participants
Arm/Group | PF-02545920 20 mg BID | PF-02545920 5 mg BID | Placebo
Number analyzed (Participants) | 87 | 95 | 88
participants | 76 (8.63) | 82 (7.30) | 63 (6.67)

4. Secondary Outcome: Number of Participants With Serious Adverse Events
Description: Adverse event (AE) was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. An serious adverse event (SAE) was an AE resulting in any of the following outcomes or deemed significant for any other reason: death, initial or prolonged inpatient hospitalization, life-threatening experience (immediate risk of dying), persistent or significant disability or incapacity, congenital anomaly.
Time Frame: Day 1, 7, 14, 28, 56, 91, 133, 182 and follow-up visits (from Day 189 to 192)
Population: All participants with at least one dose of study medication.
Measure: Number; unit: participants
Arm/Group | PF-02545920 20 mg BID | PF-02545920 5 mg BID | Placebo
Number analyzed (Participants) | 87 | 95 | 88
participants | 8 (8.63) | 2 (7.30) | 7 (6.67)

5. Secondary Outcome: Number of Participants With Laboratory Test Abnormalities (Without Regard to Baseline Abnormalities)
Description: Following parameters were analyzed for laboratory examination: hematology (hemoglobin, hematocrit, red blood cell count, platelet count, white blood cell count, total neutrophils, eosinophils, monocytes, basophils, lymphocytes);coagulation (PT international ratio); liver function (total bilirubin, direct bilirubin, indirect bilirubin, aspartate aminotransferase, alanine aminotransferase, gamma GT, LDH, alkaline phosphatase, total protein, albumin); renal function (blood urea nitrogen, creatinine, uric acid); electrolytes (calcium, sodium, potassium, chloride, total bicarbonate, magnesium, phosphate); clinical chemistry (glucose, glycosylated, hemoglobin, human chorionic gonadotropin, creatine kinase); urinalysis (decimal logarithm of reciprocal of hydrogen ion activity [pH], urine specific gravity, glucose, protein, blood, ketones, nitrite).
Time Frame: Screening, Day 1, 7, 14, 28, 56, 91, 133, 182 and follow-up visits (from Day 189 to 192)
Population: All participants with at least one dose of study medication.
Measure: Number; unit: participants
Arm/Group | PF-02545920 20 mg BID | PF-02545920 5 mg BID | Placebo
Number analyzed (Participants) | 86 | 95 | 88
participants | 47 (8.63) | 46 (7.30) | 48 (6.67)

6. Secondary Outcome: Number of Participants With Laboratory Test Abnormalities (With Normal Baseline)
Description: as for outcome 5
Time Frame: Screening, Day 1, 7, 14, 28, 56, 91, 133, 182 and follow-up visits (from Day 189 to 192)
Population: All participants with at least one dose of study medication.
Measure: Number; unit: participants
Arm/Group | PF-02545920 20 mg BID | PF-02545920 5 mg BID | Placebo
Number analyzed (Participants) | 86 | 95 | 88
participants | 40 (8.63) | 36 (7.30) | 41 (6.67)

7. Secondary Outcome: Number of Participants With Vital Sign Data That Met Criteria for Potential Clinical Concern (Absolute Values)
Description: Absolute values were analyzed for supine systolic blood pressure (SBP), standing SBP, supine diastolic blood pressure (DBP), standing DBP, supine pulse rate, and standing pulse rate. Number of participants with vital signs data meeting the following criteria was reported: Criterion A: supine SBP less than (<) 90 millimeter of mercury(mmHg); Criterion B: standing SBP < 90 mmHg; Criterion C: supine DBP <50 mmHg; Criterion D: standing DBP <50 mmHg; Criterion E: supine pulse rate < 40 beats per minute(BPM); Criterion F: supine pulse rate greater than (>)120 BPM; Criterion G: standing pulse rate < 40 beats per minute(BPM); Criterion H: standing pulse rate >120 BPM;
Time Frame: Screening, Day 1, 28, 91, and 182
Population: All participants with at least one dose of study medication.
Measure: Number; unit: participants
Arm/Group | PF-02545920 20 mg BID | PF-02545920 5 mg BID | Placebo
Number analyzed (Participants) | 87 | 95 | 88
participants
  Criterion A | 1 (8.63) | 0 (7.30) | 0 (6.67)
  Criterion B | 3 | 2 | 3
  Criterion C | 2 | 1 | 1
  Criterion D | 1 | 3 | 0
  Criterion E | 0 | 0 | 0
  Criterion F | 0 | 0 | 1
  Criterion G | 0 | 0 | 0
  Criterion H | 0 | 0 | 0

8. Secondary Outcome: Number of Participants With Vital Sign Data That Met Criteria for Potential Clinical Concern (Increase From Baseline)
Description: The number of participants with vital signs data of maximum increase from baseline meeting the following criteria was reported: Criterion A: maximum increase from baseline in supine SBP greater than or equal to (>=) 30 mmHg; Criterion B: maximum increase from baseline in standing SBP >= 30 mmHg; Criterion C: maximum increase from baseline in supine DBP >=20 mmHg; Criterion D: maximum increase from baseline in standing DBP >=20 mmHg
Time Frame: Screening, Day 1, 28, 91, and 182
Population: All participants with at least one dose of study medication.
Measure: Number; unit: participants
Arm/Group | PF-02545920 20 mg BID | PF-02545920 5 mg BID | Placebo
Number analyzed (Participants) | 87 | 95 | 88
participants
  Criterion A | 4 (8.63) | 1 (7.30) | 4 (6.67)
  Criterion B | 7 | 8 | 6
  Criterion C | 3 | 3 | 10
  Criterion D | 3 | 8 | 9

9. Secondary Outcome: Number of Participants With Vital Sign Data That Met Criteria for Potential Clinical Concern (Decrease From Baseline)
Description: The number of participants with vital signs data of maximum decrease from baseline meeting the following criteria was reported: Criterion A: maximum decrease from baseline in supine SBP >= 30 mmHg; Criterion B: maximum decrease from baseline in standing SBP >= 30 mmHg; Criterion C: maximum decrease from baseline in supine DBP >=20 mmHg; Criterion D: maximum decrease from baseline in standing DBP >=20 mmHg
Time Frame: Screening, Day 1, 28, 91, and 182
Population: All participants with at least one dose of study medication.
Measure: Number; unit: participants
Arm/Group | PF-02545920 20 mg BID | PF-02545920 5 mg BID | Placebo
Number analyzed (Participants) | 87 | 95 | 88
participants
  Criterion A | 1 (8.63) | 7 (7.30) | 3 (6.67)
  Criterion B | 9 | 8 | 9
  Criterion C | 8 | 6 | 8
  Criterion D | 10 | 14 | 9

10. Secondary Outcome: Number of Participants With Electrocardiogram (ECG) Data That Met Criteria for Potential Clinical Concern(Absolute Values)
Description: The number of participants with ECG absolute values meeting the following criteria was reported: Criterion A: maximum PR interval (time from the beginning of P wave to the start of QRS complex, corresponding to the end of atrial depolarization and onset of ventricular depolarization) >=300 msec; Criterion B: maximum QRS complex(time from Q wave to the end of S wave, corresponding to ventricle depolarization) >=140 msec; Criterion C: maximum QTcF interval (time from the beginning of Q wave to the end of T wave corresponding to electrical systole, corrected for heart rate using Fridericia's formula) 450-<480 msec; Criterion D: maximum QTcF interval 480-<500 msec; Criterion E: maximum QTcF interval (Fridericia's correction) >=500 msec
Time Frame: Screening, Day 1, 28, 91, and 182
Population: All participants with at least one dose of study medication.
Measure: Number; unit: participants
Arm/Group | PF-02545920 20 mg BID | PF-02545920 5 mg BID | Placebo
Number analyzed (Participants) | 86 | 93 | 88
participants
  Criterion A | 0 (8.63) | 0 (7.30) | 0 (6.67)
  Criterion B | 0 | 0 | 0
  Criterion C | 5 | 2 | 7
  Criterion D | 0 | 0 | 0
  Criterion E | 0 | 0 | 0

11. Secondary Outcome: Number of Participants With Electrocardiogram (ECG) Data That Met Criteria for Potential Clinical Concern(Increase From Baseline)
Description: Number of participants with ECG meeting the following criteria was reported: Criterion A: maximum PR interval increase from baseline percentage change (PctChg)>= 25/50%; Criterion B: maximum QRS complex increase from baseline PctChg >=50%; Criterion C: maximum QTcF interval (Fridericia's correction) increase from baseline 30<=change<60 msec; Criterion D: maximum QTcF interval (Fridericia's correction) increase from baseline change >=60 msec.
Time Frame: Screening, Day 1, 28, 91, and 182
Population: All participants with at least one dose of study medication.
Measure: Number; unit: participants
Arm/Group | PF-02545920 20 mg BID | PF-02545920 5 mg BID | Placebo
Number analyzed (Participants) | 86 | 93 | 88
participants
  Criterion A | 0 (8.63) | 0 (7.30) | 0 (6.67)
  Criterion B | 0 | 0 | 0
  Criterion C | 4 | 4 | 6
  Criterion D | 1 | 0 | 0

12. Secondary Outcome: Severity of Adverse Events Related to Extrapyramidal Symptoms (EPS) Including Dystonia and Akathisia
Description: Adverse event (AE) was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. AE was assessed according to severity; mild (not causing any significant problem, dose adjustment not required), moderate (caused problem that does not interfere significantly with usual activities or the clinical status, dose adjustment needed due to adverse event) and severe (caused problem that interferes significantly with usual activities or the clinical status, study drug stopped due to adverse event). EPS were reported AEs of dystonia and akathisia.
Time Frame: Day 1, 7, 14, 28, 56, 91, 133, 182 and follow-up visits (from Day 189 to 192)
Population: All participants with at least one dose of study medication.
Measure: Number; unit: participants
Arm/Group | PF-02545920 20 mg BID | PF-02545920 5 mg BID | Placebo
Number analyzed (Participants) | 87 | 95 | 88
participants
  Dystonia(Mild) | 0 (8.63) | 0 (7.30) | 0 (6.67)
  Dystonia(Moderate) | 0 | 0 | 0
  Dystonia(Severe) | 1 | 0 | 0
  Akathisia(Mild) | 1 | 2 | 0
  Akathisia(Moderate) | 2 | 1 | 0
  Akathisia(Severe) | 0 | 0 | 0

13. Secondary Outcome: Change From Baseline in the Total Maximum Chorea (TMC) Score of the UHDRS After 13 and 26 Weeks of Treatment.
Description: The UHDRS was a clinical rating scale which has been developed by the Huntington Disease Study Group (HSG) to provide a uniform assessment of the clinical features and course of HD. The components of the full UHDRS assess motor function, cognition, behavior and functional abilities. The Total Maximum Chorea (TMC) was a subset of the TMS assessment. It was composed of the scoring of 7 chorea assessments (face, orobuccolingual, trunk, right and left upper extremities, right and left lower extremities). Each assessment was rated from 0 to 4 (absent to prolonged). TMC is obtained by adding up each of the separate scores, leading to max score of 28. The minimum score is 0. The higher the score, the worse the symptoms. n is the number of evaluable subjects in each visit.
Time Frame: Baseline, Week 13, Week 26
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | PF-02545920 20 mg BID | PF-02545920 5 mg BID | Placebo
Number analyzed (Participants) | 84 | 95 | 88
units on a scale
  Week 13: number analyzed (Participants) | 67 | 83 | 77
  Week 13 | 1.1 (3.92) | -0.2 (3.50) | -0.9 (2.56)
  Week 26: number analyzed (Participants) | 59 | 83 | 80
  Week 26 | 0.7 (3.81) | -0.4 (2.84) | -0.8 (2.79)
Statistical Analysis 1: Comparison: PF-02545920 20 mg BID vs Placebo; Week 13; Test type: Superiority or Other; p = 0.0030, MMRM; Mean Difference (Net) = 1.54, 90% CI 2-sided [0.69 to 2.39], Standard Error of Mean 0.515
Statistical Analysis 2: Comparison: PF-02545920 5 mg BID vs Placebo; Week 13; Test type: Superiority or Other; p = 0.4656, MMRM; Mean Difference (Net) = 0.36, 90% CI 2-sided [-0.45 to 1.17], Standard Error of Mean 0.491
Statistical Analysis 3: Comparison: PF-02545920 20 mg BID vs Placebo; Week 26; Test type: Superiority or Other; p = 0.0149, MMRM; Mean Difference (Net) = 1.21, 90% CI 2-sided [0.39 to 2.02], Standard Error of Mean 0.492
Statistical Analysis 4: Comparison: PF-02545920 5 mg BID vs Placebo; Week 26; Test type: Superiority or Other; p = 0.8233, MMRM; Mean Difference (Net) = 0.10, 90% CI 2-sided [-0.66 to 0.86], Standard Error of Mean 0.460

14. Secondary Outcome: Number of Participants With Suicidal Ideation or Suicidal Behavior as Assessed by the Columbia Suicide Severity Rating Scale (C-SSRS) From Baseline to Follow-up Visit
Description: The C-SSRS captured the occurrence, severity, and frequency of suicide-related thoughts and behaviors during the assessment period. C-SSRS assessed whether participant experienced following: completed suicide; suicide attempt; preparatory acts towards imminent suicidal behavior; suicidal ideation; self-injurious behavior, no suicidal intent. The results presented are the number of participants with completed suicide or non-fatal suicide events or behaviors. Worsening of suicidal ideation was an increase in severity of suicidal ideation from baseline.
Time Frame: Day 1, 7, 14, 28, 56, 91, 133, 182 and follow-up visits (from Day 189 to 192)
Population: All participants with at least one dose of study medication.n is the number of evaluable participants in each visit
Measure: Number; unit: participants
Arm/Group | PF-02545920 20 mg BID | PF-02545920 5 mg BID | Placebo
Number analyzed (Participants) | 87 | 95 | 88
participants
  Completed Suicide | 0 (8.63) | 0 (7.30) | 0 (6.67)
  Suicide Attempt | 1 | 0 | 0
  Imminent Suicidal Behavior | 1 | 1 | 0
  Suicidal Ideation | 7 | 5 | 4
  Self-Injurious Behavior, No Suicidal Attempt | 1 | 0 | 0

15. Secondary Outcome: Clinical Global Impression of Improvement (CGI-I) Scale Score After 13 and 26 Weeks of Treatment.
Description: CGI-I: 7-point clinician rated scale ranging from 1 (very much improved) to 7 (very much worse). Clinician responded to a question: "Compared to your subject's condition at the beginning of treatment, how much has your subject changed?". Improvement was compared to baseline and was defined as a score of 1 (very much improved), 2 (much improved), or 3 (minimally improved) on the scale. Higher score = more affected. n is the number of evaluable participants in each visit.
Time Frame: Week 13 & Week 26
Population: All participants who have been randomized and have taken at least one dose of PF-02545920 or placebo. Participants without post-dose measurements will not contribute to the analysis, except in the description of the baseline values.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | PF-02545920 20 mg BID | PF-02545920 5 mg BID | Placebo
Number analyzed (Participants) | 84 | 95 | 88
units on a scale
  Week 13: number analyzed (Participants) | 66 | 83 | 77
  Week 13 | 4.0 (1.00) | 3.7 (0.90) | 3.6 (0.83)
  Week 26: number analyzed (Participants) | 59 | 83 | 80
  Week 26 | 3.9 (1.13) | 3.8 (0.99) | 3.8 (0.91)
Statistical Analysis 1: Comparison: PF-02545920 20 mg BID vs Placebo; Week 13; Test type: Superiority or Other; p = 0.0181, MMRM; Mean Difference (Net) = 0.35, 90% CI 2-sided [0.11 to 0.60], Standard Error of Mean 0.148
Statistical Analysis 2: Comparison: PF-02545920 5 mg BID vs Placebo; Week 13; Test type: Superiority or Other; p = 0.7133, MMRM; Mean Difference (Net) = 0.05, 90% CI 2-sided [-0.18 to 0.28], Standard Error of Mean 0.140
Statistical Analysis 3: Comparison: PF-02545920 20 mg BID vs Placebo; Week 26; Test type: Superiority or Other; p = 0.4657, MMRM; Mean Difference (Net) = 0.12, 90% CI 2-sided [-0.15 to 0.39], Standard Error of Mean 0.163
Statistical Analysis 4: Comparison: PF-02545920 5 mg BID vs Placebo; Week 26; Test type: Superiority or Other; p = 0.8339, MMRM; Mean Difference (Net) = 0.03, 90% CI 2-sided [-0.22 to 0.28], Standard Error of Mean 0.150

ADVERSE EVENTS:
Time Frame: Day 1, 7, 14, 28, 56, 91, 133, 182 and follow-up visits (from Day 189 to 192)
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one participant and as non-serious in another participant, or one participant may have experienced both a serious and non-serious event during the study.
Arm/Group | PF-02545920 5 mg BID | Placebo | PF-02545920 20 mg BID
Serious Adverse Events (participants affected / at risk) | 2/95 | 7/88 | 8/87
Other Adverse Events (participants affected / at risk) | 71/95 | 42/88 | 65/87
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | PF-02545920 5 mg BID (N=95) | Placebo (N=88) | PF-02545920 20 mg BID (N=87)
Atrial fibrillation (Cardiac disorders) | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 0
General physical health deterioration (General disorders) | 0 | 0 | 2
Clostridium difficile colitis (Infections and infestations) | 0 | 1 | 0
Pneumonia (Infections and infestations) | 0 | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 1 | 0
Head injury (Injury, poisoning and procedural complications) | 0 | 1 | 0
Rib fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Weight decreased (Investigations) | 0 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Syncope (Nervous system disorders) | 0 | 0 | 1
Vestibular migraine (Nervous system disorders) | 0 | 1 | 0
Device occlusion (Product Issues) | 0 | 0 | 1
Acute stress disorder (Psychiatric disorders) | 0 | 1 | 0
Agitation (Psychiatric disorders) | 1 | 0 | 0
Anxiety (Psychiatric disorders) | 1 | 1 | 0
Major depression (Psychiatric disorders) | 0 | 0 | 2
Suicidal behaviour (Psychiatric disorders) | 0 | 0 | 1
Suicidal ideation (Psychiatric disorders) | 0 | 1 | 1
Suicide attempt (Psychiatric disorders) | 0 | 0 | 1
Asphyxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | PF-02545920 5 mg BID (N=95) | Placebo (N=88) | PF-02545920 20 mg BID (N=87)
Diarrhoea (Gastrointestinal disorders) | 7 | 6 | 7
Dry mouth (Gastrointestinal disorders) | 1 | 0 | 6
Nausea (Gastrointestinal disorders) | 12 | 7 | 11
Vomiting (Gastrointestinal disorders) | 10 | 3 | 7
Fatigue (General disorders) | 11 | 9 | 16
Nasopharyngitis (Infections and infestations) | 18 | 12 | 8
Urinary tract infection (Infections and infestations) | 5 | 3 | 4
Fall (Injury, poisoning and procedural complications) | 15 | 9 | 5
Weight decreased (Investigations) | 6 | 1 | 15
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 | 5 | 2
Chorea (Nervous system disorders) | 4 | 1 | 8
Dizziness (Nervous system disorders) | 1 | 4 | 10
Dyskinesia (Nervous system disorders) | 0 | 1 | 9
Headache (Nervous system disorders) | 8 | 8 | 8
Sedation (Nervous system disorders) | 5 | 0 | 2
Somnolence (Nervous system disorders) | 9 | 3 | 16
Anxiety (Psychiatric disorders) | 6 | 2 | 12
Insomnia (Psychiatric disorders) | 4 | 2 | 11
Irritability (Psychiatric disorders) | 7 | 1 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.